CLINICAL TRIAL: NCT01125462
Title: Post Marketing Assessment of GONAL-f Solution for Injection in a Prefilled Pen for Follicular Stimulation in IVF-ET Cycles: An Observational Study
Brief Title: A Post Marketing Assessment of Gonal f Solution for Injection in a Prefilled Pen for Follicular Stimulation in in Vitro Fertilisation/Embryo Transfer (IVF-ET) Cycles
Acronym: POINT
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck d.o.o., Serbia (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 700623-517
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Infertility
Keywords: Ovulation Induction; Infertility; Gonal-f; FertiQoL; Quality of Life
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma

GROUPS / COHORTS (2):
- Subjects previously treated with Gonal-f: Subjects who had undergone at least one treatment cycle with Gonal-f powder and solvent for solution for injection within the past 12 months (equivalent to 75 IU/ml, 450 IU/0.75ml or 1050 IU/1.75 ml)
  Interventions: Other: Quality of Life Questionnaire (FertiQoL)
- Subjects previously treated with urine-derived FSH: Subjects which had undergone at least one treatment cycle with urine-derived FSH therapy with vials within the past 12 months
  Interventions: Other: Quality of Life Questionnaire (FertiQoL)

INTERVENTIONS:
Other: Quality of Life Questionnaire (FertiQoL) — Subjects will be administered the first internationally validated Quality of Life questionnaire (FertiQoL) to assess the quality of life of infertile subjects.
  Other Names: FertiQoL

SUMMARY:
The development of recombinant DNA technology, culminated in the introduction of the first recombinant human follicle stimulating hormone (r hFSH), Gonal-f, which further developed to become Gonal-f Filled-by-Mass (FbM) pen has been used in the fertility treatment since many years. It has been found that subjects using the pen found it less stressful, easier to use and more convenient than a conventional syringe and would recommend the prefilled pen to another woman considering gonadotropin treatment. However, the use of the Gonal-f (FbM) pen between Serbian subjects is on a very low level though the Gonal f vials with the 75 IU of follitropin alfa have been present in Serbian market since 2003. On the contrary from the clinical practice in European countries, Serbian subjects usually receive daily dose of injectable gonadotropins at the IVF clinics or by partner/family member.

This open-label, multicentric, observational non-interventional study is designed with the aim to know the reason of Serbian subjects not injecting themselves with Gonal f and the quality of life (QoL) of Serbian women/couples with the infertility problem.

DETAILED DESCRIPTION:
Fertility is the ability to conceive or induce conception. A normal fertile couple has about a 20% chance of achieving pregnancy in any one month of unprotected intercourse. Infertility is defined as the failure to conceive after 12 months of unprotected intercourse. It is generally estimated that about 10% to 15% of couples can be classified as having conception difficulties. About 30% of these are as a result of female factors, 30% as a result of male factors and a further 30% are due to a combination of both male and female factors. In about 10% of cases, the underlying cause is not found (unexplained fertility).

Follicle-stimulating hormone is one of the key hormones regulating reproductive functions both in females and males. In females, it stimulates the development of ovarian follicles which carry the oocytes, while in males it promotes spermatogenesis. Follicle-stimulating hormone binding to its receptor triggers intracellular mechanisms that regulate steroidogenesis, cell replication and expression of specific proteins and growth that modulate gametogenesis. Complete or partial deficiencies in FSH secretion are common causes of infertility in both women and men. Administration of FSH, either alone or in combination with luteinizing hormone (LH), has been used successfully to treat these infertility problems. Nearly 40% of women who are infertile have an ovulatory problem. These disorders may originate in the pituitary, the hypothalamus, the ovaries, or the anatomy of the reproductive system.

Over the last 50 years the quality of FSH used in fertility treatment for inducing follicular development has improved via several distinguishable steps. For many years only human menopausal gonadotropin (hMG), a mixture of human LH and FSH extracted from the urine of post-menopausal women, was available for treatment of infertility. However, Merck Serono has developed the recombinant human FSH (r-hFSH) for clinical use, which has been in the market for several years. This development has been guided by the quest for control over the variability in urinary derived drugs. The recombinant system is a well-defined and controlled manufacturing process, which means that the content of these recombinant gonadotropins is consistent from batch-to-batch, accurately measured and filled-by-mass (i.e. in terms of weight in micrograms). This allows precise dosing control in both ovulation induction (OI) and assisted reproduction techniques (ART). Recombinant human fertility hormones are considered to have consistency of the source material and of the active product, the purity and specific activity of the protein, a good efficacy, safety and tolerability.

OBJECTIVES

Primary objective:

* To evaluate the ease-of-use of Gonal-f (FbM) in a prefilled pen in normal clinical practice conditions under different protocols of follicular stimulation

Secondary objective:

* To evaluate the local tolerability (incidence of local reaction at the injection site) to drug administration.

This study is planned to be conducted in 3 IVF/ART clinics in Serbia recruiting approximately 20 subjects per centre (10 to each group) giving a total of 60 subjects. Subjects with previous stimulation treatment by the use of some injectable gonadotropins and not the stimulation with clomiphene citrate will be enrolled in this study. Depending on the kind of gonadotropin used in the previous stimulation treatment the subject has been treated with (meaning either Gonal-f ampules or urinary derived drugs), subjects will be stratified into two groups. The first group will include subjects who have undergone at least one treatment cycle with Gonal f powder and solvent for solution for injection within the past 12 months (equivalent to 75 IU/ml, 450 IU/0.75ml or 1050 IU/1.75 ml). The second group will include subjects which had undergone at least one treatment cycle with urine-derived FSH therapy with vials within the past 12 months. Subjects in both groups included in the study will be treated according to the Summary of Product Characteristics (SmPC) and according to clinical practice at each site. These subjects will also answer on questions from the first internationally validated QoL questionnaire called FertiQoL. The FertiQoL is the instrument that surveys infertile subjects to assess their QoL. Each and every subject will undergo one stimulation treatment cycle and each subject should be followed for approximately 2 weeks or until chemically proven pregnancy. After treatment, subject satisfaction with the Gonal f (FbM) prefilled pen will be measured using a post-treatment questionnaire in which participants will be asked to compare their treatment experiences and choose a preferred injection method.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing superovulation prior to assisted reproductive techniques such as IVF
* Subjects who have given written informed consent with the understanding that consent may be withdrawn by the subject at any time without prejudice for her future medical care
* Female subjects between 18-43 years of age who have undergone at least one treatment cycle and as such are not included in the fertility reimbursed program supported by Serbian Ministry of Health
* Subjects willing and able to comply with the protocol for the duration of the study
* Subjects who have early follicular phase (day 2-4) serum level of basal FSH lower and equal to 12 IU/L measured in the centre's local laboratory (i.e. within 2 months prior to inclusion).
* If subject is supposed to gone through ovarian induction (OI), criteria for inclusion in the study is to receive the treatment with the Gonal f (FbM) Prefilled Pen for at least 5-6 days

Exclusion Criteria:

* Subjects with ovarian, uterine or mammary cancer
* Pregnancy and lactation period
* Subjects with tumours of the hypothalamus and pituitary gland
* Subjects with uterine myoma requiring treatment
* Subjects with ovarian enlargement or cyst of unknown aetiology
* Subjects with a clinically significant systemic disease
* Subjects with abnormal gynaecological bleeding of undetermined origin
* Subjects with known allergy or hypersensitivity to human gonadotropin preparations
* Subjects who have entered previously into this study or simultaneous participation in another study
* Subjects with legal incapacity or limited legal capacity

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pre-menopausal woman, between 18-43 years old requiring treatment with recombinant FSH for controlled ovarian hyperstimulation for IVF or OI in Serbia
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who preferred the Gonal-f (FbM) Pen to vials | Post-treatment with Gonal-f (2 weeks after embryo transfer)

SECONDARY OUTCOMES:
Assessment of effectiveness of Gonal-f | One stimulation treatment cycle until 7 weeks of intrauterine pregnancy or mensuration
  Total dose of r-hFSH used during the stimulation period, number of days of stimulation treatment, cancellation rates (not administring hCG due to poor response to stimulation), total number of retrieved oocytes (34-36 hours after hCG administration), mean number of embryos transferred, embryo implantation rate, number of miscarriages, registration of body mass index (BMI), registration of smoking habit (previous or present)
Local tolerance of Gonal-f (FbM) solution for injection in a prefilled pen | Screening period to post-treatment with Gonal-f (until 7 weeks of intrauterine pregnancy)
  Local tolerance of Gonal-f (FbM) solution for injection in a prefilled pen (pain, bruising, redness, itching, swelling as documented by the subject) and adverse events encountered during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jasmina Cvetkovic, PhD, Study Director — Merck d.o.o., Serbia
Locations (3):
- Serbia (3):
  - Dept. for Human Reproduction, Clinical Centre Vojvodina, Novi Sad, Branimira Ćosića 37
  - University hospital for Gynaecology and Obstetrics "Narodni front", Dept. for ART, Belgrade, Kraljice Marije 62
  - Clinical Centre Serbia, Visegradska, Belgrade